CLINICAL TRIAL: NCT03956563
Title: Effect of Hybrid Laser 10600+1540 nm on Vaginal Atrophy-genitourinary Syndrome of the Menopause
Brief Title: Effect of Hybrid Laser 10600+1540 nm on GSM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Quanta System, S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YLMT_VAG
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Vaginal Atrophy; Genitourinary Disease
MeSH Terms: conditions — Urogenital Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment arm (Active Comparator): Youlaser MT: sequential 10600+1540 nm with vaginal (2 passes) and intritus (1 pass) treatment
  Interventions: Device: Youlaser MT Group 1
- Control arm (Sham Comparator): Youlaser MT: no laser emission with vaginal (2 passes) and intritus (1 pass) treatment
  Interventions: Device: Youlaser MT Group 2

INTERVENTIONS:
Device: Youlaser MT Group 2 — Youlaser MT is a laser device including two laser sources emitting at 10600 nm (CO2) and 1540 nm (Ga-As) intended to be used for gynaecological applications.
  Each patient in the control arm will receive 3 simulated laser treatments every 30 days.
  A placebo consists in a sham device laser that simulates the acoustic signal even if it does not deliver any laser radiation to the subject.
  Arms: Control arm
Device: Youlaser MT Group 1 — Youlaser MT is a laser device including two laser sources emitting at 10600 nm (CO2) and 1540 nm (Ga-As) intended to be used for gynaecological applications.
  Each patient in the active arm will receive 3 laser treatments with the laser: one treatment administration every 30 days.
  Arms: Active treatment arm

SUMMARY:
The primary objective of the study is to clinically confirm, by comparison with a control group, the performance of the 10600 +1540 nm laser in the improvement of atrophic vaginal epithelium at 3 months after the last laser treatment.

The secondary objectives are:

1. Confirm the performance of 10600 +1540 nm laser in the improvement of atrophic vaginal epithelium at 9 months post-laser treatment, and compare it with the results at 3 months.
2. Evaluate the improvement of the GSM urinary symptoms and urinary incontinence (UI) and their impact on the Quality of Life, at each timepoint after the first laser treatment.
3. To assess the Patient's Global Impression of Improvement (PGI) with the laser treatment

   * For the GSM symptoms
   * For the urinary symptoms and UI
4. To assess the patient's satisfaction with the laser treatment.

   * For the GSM symptoms
   * For the urinary symptoms and UI.

ELIGIBILITY:
Inclusion Criteria:

1. Menopausal women (defined as ³1 year without menstruation until 65 years of age and no more than 10 years within the menopause) with at least 1 GSM symptom (vaginal dryness, burning, itching or dyspareunia ) Atrophic vaginal epithelium measured with the VMV values of 0-49%
2. To have any of the urinary symptoms: urgency, frequency, nocturia and urinary incontinence as symptoms of GSM
3. Women able to understand , accept and signed the Informed Consent.
4. Women with adequate physical and mental ability to understand and complete the questionnaires of quality of life and with cooperative attitude.

Exclusion Criteria:

1. VMV 50-64% (moderate) 65-100% (high estrogenic effect on the vaginal epithelium)
2. Impossibility of introducing the laser device
3. History or other energy-based vaginal therapy within 6 months prior to enrollment.
4. Being on hormone replacement therapy to relieve menopausal symptoms 3 months before the study.
5. Being on regular and effective topical estrogen therapy within the last 3 months.
6. Being on concomitant anticoagulants therapy .
7. Patients suffering of epileptic attacks and immunosuppressive diseases.
8. Daily and effective use of moisturizers, lubricants or probiotics.
9. Previous pelvic radiotherapy or brachytherapy
10. Gynecologic or rectal cancer less than 5 years ago
11. Breast cancer with antiestrogenic therapy
12. Bladder emptying dysfunction.
13. Women operated on UI.
14. Subjects undergoing conservative supervised treatment, such as pelvic floor rehabilitation exercises.
15. Genital prolapse grade III or higher, according to the simplified POPQ classification.
16. Being on effective pharmacological treatment for overactive bladder.
17. Taking diuretics.
18. Patients with neurological diseases (Multiple Sclerosis, spinal cord injury, stroke, Parkinson's)
19. Insulin-dependent diabetes mellitus (IDDM) or non-dependent insulin poorly controlled.
20. Body Mass Index (BMI) > 40 kg/m2
21. Active urinary tract infection
22. Hematuria.
23. Women who present active or recurrent genital herpes.
24. Undiagnosed metrorrhagia
25. Abnormal last cervical cytology
26. Developmental disability, cognitive impairment and/or serious mental health illness.
27. Language barrier.
28. Women who refuse to participate in the study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
Atrophic vaginal epithelium change | 3 months and 9 months post laser treatments
  The primary efficacy outcome measure in this study is to obtain on the atrophic vaginal epithelium at 3 months after the last laser treatment, values going from absent/low estrogenization (0-49%) to moderate or high estrogenization (50-64%) measured with VMV. The results will be compared between the treatment and the control arm.

SECONDARY OUTCOMES:
Treatment area success for GSM #1 | 3 months and 9 months post laser treatments
  Change to vaginal pH<5
Treatment area success for GSM #2 | 3 months and 9 months post laser treatments
  Decrease in the GSM symptoms on VAS scale 0-10. vaginal dryness, burning, itching, and dyspareunia,dysuria (0: complete absence of symptoms, 10: worst possible symptoms).
Treatment area success for Urinary incontinence #1 | 3 months and 9 months post laser treatments
  Change in ICIQ-SF score from moderate to mild incontinence, or from mild to nil incontinence.
  Improve the quality of life related to incontinence by decreasing the score in the interference with everydays life question.
Treatment area success for Urinary incontinence #2 | 3 months and 9 months post laser treatments
  Change in Sandvick test score from moderate to mild incontinence, or from mild to nil incontinence.
Treatment area success for Urinary incontinence #3 | 3 months and 9 months post laser treatments
  Decrease in the GSM urinary symptoms for dysuria and nocturia on VAS sclae 0-10
Patient Global Impression | 3 months and 9 months post laser treatments
  Score in the Patient Global Impression of Improvement, as better and much better.
Patient Satisfaction | 3 months and 9 months post laser treatments
  Score in the degree of patient satisfaction, as satisfied and very satisfied.
Safety evaluation | 61 days (at each treatment)
  Each of the following safety outcome variables recorded across study duration will be assessed
  1. Pain rating during and after laser treatment.
  2. Frequence and severity of potential adverse effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrician & Gynecologist Hospital Universitario Sant Joan de Reus, Reus, Spain

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601